CLINICAL TRIAL: NCT00922610
Title: An Open-label Study of the Effect of Mircera on Hemoglobin Levels in Filipino Chronic Kidney Disease Patients
Brief Title: A Study of Mircera in Renal Anemia Among Filipino Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21983
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — sc every 2 weeks at a starting dose of 0.6micrograms/kg;subsequently every 4 weeks

SUMMARY:
This study will assess the efficacy and safety of once monthly administration of Mircera in Filipino patients with chronic kidney disease who are either on dialysis or predialysis, and not receiving erythropoiesis stimulating agents.Patients will receive Mircera at a starting dose of 0.6 micrograms/kg sc every 2 weeks, with dose adjustments until a target hemoglobin level is achieved, and then dosing will continue every 4 weeks. The anticipated time on study treatment is 3-12 months, and the target sample is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic kidney disease;
* anemia (Hb >8 and <11 g/dL);
* regular dialysis or predialysis, not treated with ESA.

Exclusion Criteria:

* transfusion of red blood cells during previous 8 weeks;
* poorly controlled hypertension;
* overt gastrointestinal bleeding, or other bleeding necessitating transfusion during previous 8 weeks;
* active malignant disease (except melanoma of skin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Increase in Hb >1.0g/dL from baseline, and Hb conc. >11g/dL without red blood cell transfusion, for dialysis patients;Hb conc >11-12 g/dL for pre-dialysis patients | 24 weeks after first dose, through week 25

SECONDARY OUTCOMES:
>=60% responders with target Hb >11g/dL for dialysis patients; Hb conc >11-12g/dL for pre-dialysis patients;incidence of RBC transfusions; no. of patients with dose adjustments | At end of 24 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Philippines (5):
  - Cavite
  - Makati City
  - Manila
  - Marikina City
  - Pasig